CLINICAL TRIAL: NCT05299944
Title: Reducing Pain and Opioid Use With CBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-5122
Record Dates: First submitted 2022-02-22; First posted 2022-03-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
Keywords: Opioids; Pain; Cannabidiol; CBD; Cannabis
MeSH Terms: conditions — Opioid-Related Disorders; Pain; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full-spectrum Cannabidiol (Active Comparator): 210mg/day of full-spectrum cannabidiol, containing less than 0.3%THC.
  Interventions: Drug: Cannabidiol
- Broad-spectrum Cannabidiol (Active Comparator): 210mg/day of broad-spectrum cannabidiol, containing 0%THC.
  Interventions: Drug: Cannabidiol
- Hemp Seed Oil Placebo (Placebo Comparator): 210mg/day of hemp-seed oil with no cannabinoids present.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The current study will directly test the hypothesis that a moderate dose of CBD leads to a reduction in opioid consumption, opioid craving, pain, peripheral markers of inflammation, and anxiety, as well as changes in sleep, AEA, and cognition.
  Other Names: CBD
  Arms: Broad-spectrum Cannabidiol; Full-spectrum Cannabidiol
Drug: Placebo — Placebo arm
  Arms: Hemp Seed Oil Placebo

SUMMARY:
This is a double-blind, placebo-controlled, parallel group study designed to assess the tolerability and efficacy of fsCBD and bsCBD, compared to a placebo control, to reduce opioid use, anxiety, and pain and improve sleep and cognitive function. If eligible for the study, subjects will be randomized to receive one of the conditions for 12 weeks.

DETAILED DESCRIPTION:
To better understand the effects of hemp-derived CBD with and without a small amount of THC, the investigators propose a Phase II randomized clinical trial (RCT) to examine the safety, tolerability, and clinical effects of Full Spectrum CBD (fsCBD, contains less than 0.3% THC) vs. Broad Spectrum CBD (bsCBD, does not contain THC), vs. a matching placebo in a population of opioid users.

This is a double-blind, placebo-controlled, parallel group study designed to assess the tolerability and efficacy of fsCBD and bsCBD, compared to a placebo control, to reduce opioid use, anxiety, and pain and improve sleep and cognitive function. If eligible for the study, subjects will be randomized to receive one of the conditions for 12 weeks.

Study visits will take place both in-person and via Zoom/online. Study participants will attend four in-person visits at the University of Colorado Anschutz at Week 0 (Baseline Medical Director Screen and Medication Dispense), Week 6, and Week 12. Research staff will meet with participants over Zoom during their Week 1 visit and will be contacted weekly during the 12-week study period. Following the Week 1 Zoom visit, participants will have the option to receive the survey link via email for Weeks 2-5 and 7-11 in lieu of meeting with a research team member over Zoom to allow more flexibility in time to complete the study surveys (participants can complete surveys at their convenience within a 3-business day period). In Week 16, approximately 4 weeks after the end of dosing, a final follow-up Zoom interview will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported desire or intent to use cannabidiol to reduce pain and/or opioid use
2. Must be 18 years of age or older.

Exclusion Criteria:

1. Self-reported recreational drug use (other than opioids) in the past 30 days or failed urine screen for cocaine, benzodiazepines (if not prescribed), MDMA, sedatives, or methamphetamine;
2. Self-reported current moderate/severe alcohol use, or severe opioid use disorder on the DSM V (unless patient is medically stable and approved by personal physician as well as the Medical Director for the study);
3. Actively seeking or in treatment for or history of any substance use disorder, other than opioid use disorder;
4. Currently being treated for or diagnosed with a moderate, severe, or unstable medical illness (e.g., renal disease, liver disease, cardiovascular disease). If the person has had a recent operation, they must be cleared for study participation by their surgeon or primary care doctor. Study inclusion/exclusion will be evaluated by our medical director when there are questions about applying criteria;
5. Currently taking any of the following medications:

   1. Those known to have a major interaction with Epidiolex (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, and/or teriflunomide)
   2. Acute treatment with any antiepileptic medications (e.g. clobazam, sodium valproate)
6. Report being treated for bipolar disorder, schizophrenia, dissociative disorders, eating disorders, or any other psychotic or organic mental disorder in the last year.
7. Females of childbearing potential who are pregnant, nursing, or who are not using a reliable form of birth control.
8. Endorsing item 2 on the C-SSRS measure of suicide risk.
9. Currently using CBD for medical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Reduction in pain medication use | 0-12 Weeks
  The Time Line Follow Back is a calendar-assisted measure that can be used to assess pain medication use. The investigators will use this measure to create the pain medication use variable. For opioids users, changes in opioid use will be assessed. For non-opioid users, non-opioid pain medication will be assessed.
Reduction in THC use | 0-12 Weeks
  The Timeline Follow-back will be used to quantify and frequency of THC use.
Reduction in pain | 0-12 Weeks
  -The PROMIS Numeric Rating Scale v1.0 - Pain Intensity - 1a will be used to measure pain intensity with a one question item over the past 7 days. Higher scores indicate more pain. The PROMIS Short Form v1.1 - Pain Interference - 6b rates pain on a scale from 1 (not at all) to 5 (very much), as it refers to the degree to which pain limits or interferes with subjects' physical, mental, and social activities. Higher scores indicate greater pain interference.

SECONDARY OUTCOMES:
Change in opioid craving | 0-6 Weeks, 6-12 Weeks, 0-12 Weeks, 0-16 Weeks
  The Opioid Craving Scale will be used to assess changes in craving over time. This scale has three questions assessed using a 10-pt likert scale. Higher scores (0-30) indicate greater opioid craving.
Change in inflammation | 0-6 Weeks, 6-12 Weeks, 0-12 Weeks, 0-16 Weeks
  Differences in inflammatory markers (e.g. IL-6) will be assessed over time as a moderating factor.
Change in Anandamide (AEA) | 0-6 Weeks, 6-12 Weeks, 0-12 Weeks, 0-16 Weeks
  Differences in AEA will be assessed over time as a moderating factor.
Change in quality of life | 0-6 Weeks, 6-12 Weeks, 0-12 Weeks, 0-16 Weeks
  Changes in subjective quality of life will be assessed using the PROMIS Global-10 Short Form). Scores range from 10-50, with higher scores indicating poorer quality of life.
Change in self-reported cognitive function | 0-6 Weeks, 6-12 Weeks, 0-12 Weeks, 0-16 Weeks
  Changes in self-reported cognitive function will be assessed using the FACT-Cog. There are 37 questions on a 5-pt likert scale with higher scores indicating poorer cognition.
Reduction in anxiety | 0-12 Weeks
  The Depression Anxiety Stress Scale measures the severity of anxiety symptoms. Possible scores range from 0 to 41 with higher scores indicating a worse outcome/more severe symptoms of anxiety.
Reduction in sleep disturbance / fatigue | 0-12 Weeks
  * The PROMIS Short Form v1.0 - Sleep Disturbance - 4A measure the severity of sleep disturbances. Possible scores range from 0 to 4 with lower scores indicating a worse outcome/more severe symptoms of sleep disturbance/fatigue.
  * The PROMIS Short Form v1.0 - Fatigue - 4a measures subject fatigue over the past 7 days on a 4 point scale, with higher scores indicating more fatigue.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado - Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado